CLINICAL TRIAL: NCT02204553
Title: An Expanded Treatment Protocol of Panobinostat (LBH589) in Combination With Bortezomib and Dexamethasone in Patients With Multiple Myeloma Who Have Had at Least One Prior Line of Therapy
Brief Title: Expanded Treatment Prot of Panobinostat in Combo w/ Bortez and Dex in Pts w/ Relapsed and/or Refractory Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLBH589DUS94X
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Panobinostat; LBH589; Expanded Access; EAP, ETP; Expanded Treatment; Bortezomib; HDAC; histone deacetylace inhibitor
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Treating patients with relapsed and/or refractory Multiple Myeloma

SUMMARY:
This will be a multi-center, open label, expanded treatment protocol of panobinostat, bortezomib and dexamethasone in patients with relapsed and/or refractory multiple myeloma. Panobinostat will be administered at a starting dose of 20mg orally three times a week (every other day) for two weeks on and one week off, with dose adjustments permitted based on observed toxicity. Bortezomib will be administered either intravenously or sub-cutaneously, twice a week on days 1 and 4, two weeks on 1 week off. After 8 cycles of treatment, patients who have achieved stable disease or better by modified EBMT 1998 criteria may continue combination therapy with bortezomib dosing changed to days 1 and 8 of a 21 day cycle for up to 48 weeks of therapy. At the end of the treatment period, (48 weeks) patients with stable disease or better may continue on therapy at the discretion of their investigator until September 2015 or until drug is commercially available, whichever comes first. Patients who have not achieved at least stable disease by 8 cycles must discontinue from study treatment. Dexamethasone will be administered on the day of and the day immediately following bortezomib treatment. Patients will not receive any study treatment during the third week of each cycle. Cycles will be defined as 21 days of treatment. Investigators may not add any other anti-myeloma agents (with the exception of bisphosphonates) while patients remain on study treatment. Patients will remain on study until disease progression, unacceptable toxicity, or end of the study

ELIGIBILITY:
Inclusion Criteria:

* This study is intended for patients with relapsed and/or refractory multiple myeloma, who have received at least one prior line of therapy. Patients must require retreatment as per IMWG definitions (Kyle et al 2003). Approximately 50-100 patients are expected to be enrolled into this trial.
* Patient has a previous diagnosis of multiple myeloma, based on IMWG 2003 definitions all three of the following criteria had been met:
* Monoclonal immunoglobulin (M component) on electrophoresis, and on immunofixation on serum or on total 24 hour urine (or demonstration of M protein in cytoplasm of plasma cell for non secretory myeloma).
* Bone marrow (clonal) plasma cells ≥ 10% or biopsy proven plasmacytoma
* Related organ or tissue impairment (CRAB symptoms: anemia, hypercalcemia, lytic bone lesions, renal insufficiency, hyperviscosity, amyloidosis or recurrent infections)
* Patients who have received allogeneic stem cell transplant and do not have active graft vs host disease requiring immunosuppressive therapy are eligible.
* Patient with multiple myeloma (per IMWG 2003 definition) that is relapsed and/or refractory to at least one prior line of therapy and requires retreatment
* Relapsed-and-refractory to a therapy, provided that the patient meets any of the following conditions:
* Relapsed, defined by disease that recurred in a patient that responded under a prior therapy, by reaching a MR or better, and had not progressed under this therapy nor up to 60 days of last dose of this therapy. Patients who previously responded to treatment with BTZ are eligible.
* Patient has relapsed to at least one prior line and patient was refractory to at least one prior line by either not reaching a MR, or progressed while under this therapy, or within 60 days of its last dose. Patients previously refractory to BTZ are also eligible.
* Patients with primary refractory disease are eligible.
* Patients who have previously received high dose therapy/autologous stem cell transplant are eligible
* Patients who have received allogeneic stem cell transplant and do not have active graft vs host disease requiring immunosuppressive therapy are eligible

Exclusion Criteria:

* Patient has shown intolerance to bortezomib, dexamethasone or panobinostat or has any contraindications to any of these therapies. following available prescribing information
* Allogeneic stem cell transplant recipient presenting with graft versus host disease either active or requiring immunosuppression
* Patient has grade ≥ 2 peripheral neuropathy or grade 1 peripheral neuropathy with pain on clinical examination within 14 days of treatment
* Patient taking any anti-cancer therapy concomitantly
* Patient has second primary malignancy < 3 years of first dose of study treatment (except for treated basal or squamous cell carcinoma, or in situ cancer of the cervix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (27):
  - Ironwood Cancer and Research Centers Ironwood Cancer, Chandler, Arizona
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - Kaiser Permanente Medical Group Kaiser Permanente-Moanalua M.C, Anaheim, California
  - Alta Bates Cancer Center, Berkeley, California
  - Los Angeles Hematology/Oncology Medical Group, Los Angeles, California
  - Stanford Cancer Center Stanford Cancer Institute (2), Stanford, California
  - George Washington U Medical Center Medical Faculty Associates, Washington D.C., District of Columbia
  - University Cancer Institute Univ. Cancer Institute, Boyton Beach, Florida
  - Memorial Cancer Institute Memorial Cancer Inst., Hollywod, Florida
  - Lakes Research SC, Miami Lakes, Florida
  - Emory University School of Medicine/Winship Cancer Institute Winship Cancer Institute (2), Atlanta, Georgia
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - Hematology Oncology Clinic Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Sinai Hospital of Baltimore Sinai Hospital, Baltimore, Baltimore, Maryland
  - Bronson Battle Creek Cancer Care Center, Battle Creek, Michigan
  - University of Mississippi Medical Center Cancer Institute, Jackson, Mississippi
  - Research Medical Center Research Med. Center, Kansas City, Missouri
  - Oncology Hematology West, PC Nebraska Cancer Specialists, Omaha, Nebraska
  - Hematology Oncology of Central New Jersey, Little Silver, New Jersey
  - Morton Coleman, MD M. Coleman, MD (2), New York, New York
  - Cancer Centers of the Carolinas GHS Cancer Institute, Greenville, South Carolina
  - Wellmont Medical Associates, Bristol, Tennessee
  - Texas Oncology Texas Oncology - Arlington, Dallas, Texas
  - Texas Oncology TX Oncology Baylor, Dallas, Texas
  - Northern Utah Cancer Associates SC, Ogden, Utah
  - Virginia Oncology Associates Virginia Oncology Assoc. (2), Norfolk, Virginia
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin